CLINICAL TRIAL: NCT03937050
Title: Gestational Diabetes in Uganda and India: Design and Evaluation of Educational Films for Improving Screening and Self-management
Brief Title: Gestational Diabetes in Uganda and India Improving Screening and Self-management
Acronym: GUIDES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Indian Institute of Public Health, India (Other); Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 108-KEP-179
Record Dates: First submitted 2019-05-01; First posted 2019-05-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Gestational Diabetes
Keywords: pregnancy; gestational diabetes; India; Uganda; cluster randomized trial
MeSH Terms: conditions — Diabetes, Gestational | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): A package of three interconnected educational/behavioural film-based interventions will developed for delivery at the cluster (clinic) level. The aim of the three components will be as follows: a) improving knowledge of GDM guidelines and skills among health providers involved in GDM management, b) raising awareness of GDM and the importance of screening among pregnant women and their family members, and c) improving confidence and skills in self-management of GDM among women diagnosed.
  Interventions: Behavioral: Intervention
- Control (No Intervention): Usual care practices.

INTERVENTIONS:
Behavioral: Intervention — Three film-based components:
  1. Professional development of doctors and nurses to improve screening and management of GDM. Modules will cover knowledge and relevant clinical guidelines, skills for glucose monitoring and managing medication, specialist obstetric care, and lifestyle counselling. The films will be screened at professional development meetings.
  2. Awareness-raising among pregnant women and family members regarding GDM and the importance of healthy lifestyles during pregnancy. The film will be culturally tailored and will be screened in waiting areas of antenatal clinics/electronic versions of the films will be made available for viewing on mobile devices.
  3. Structured diabetes self-management programme for women with GDM to empower them with the necessary knowledge, skills, and confidence to manage GDM successfully. The programme will incorporate behavioural counselling and educational reinforcement. Films will be screened at group sessions/viewed on mobile devices.
  Arms: Intervention

SUMMARY:
This trial will evaluate a package of three interconnected educational/behavioural interventions aimed at: a) improving knowledge and skills of GDM guidelines and skills of health providers; b) raising awareness of importance of GDM screening among pregnant women and their families; and c) improving confidence and skills in self-management among those diagnosed with GDM. The interventions will be delivered through the medium of film as they are low-cost and scalable, and are particularly suitable for people who are not very literate, making them ideal for low- and middle-income countries (LMICs).

The research will be carried out in Uganda (Entebbe) and India (Bengaluru). A careful contextual analysis will precede the development of a culturally-tailored film-based intervention for each setting, which will be iteratively refined using qualitative research methods till it is fit for purpose. The effectiveness of the intervention will be evaluated in independent cluster randomised trials, involving ~10,000 pregnant women across 30 maternity units at each site. The films will be made available in the intervention arm facilities: for viewing by doctors and nurses at their meetings, for continual screening in waiting areas of antenatal clinics, and during group education sessions (and personal mobile use) for GDM patients. Where video/projection facilities are unavailable, small low-cost projectors will be made available. Control arms will follow usual care practices.

The principal research question is whether a low-cost educational/behavioural intervention delivered through a package of culturally-tailored films can provide scalable improvements in timely detection and management of GDM. This will be evaluated through assessing three endpoints: a) detection of GDM at 32 weeks of; b) glycaemic control (fasting glucose) in women with GDM at ~34 weeks of pregnancy; and c) adverse perinatal outcomes associated with GDM. Interviews will be conducted with women and health providers to help understand how and why the intervention may be (or may not be) successful. The ultimate aim of the project is to contribute to scientific evidence underpinning the use of films in cost-effectively scaling up behavioural interventions in low literacy settings.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18 or over attending for antenatal care at participating health facilities.
* Pregnant women willing and able to give informed consent.

Exclusion Criteria:

* Pregnant women <18 years
* No informed consent

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16500 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
GDM screening | 32 weeks of pregnancy
  Proportion of women who were tested for GDM at or after 24 weeks of pregnancy. Self-reported via telephone contact.
Mean fasting blood sugar (women with GDM) | 34 weeks of pregnancy
  Mean fasting blood sugar in women diagnosed with GDM. Measured at clinic visit.

SECONDARY OUTCOMES:
Adverse perinatal outcomes (composite measure) | 28 days postpartum (measured 6 weeks after expected date of delivery (EDD))
  Proportion of women with adverse perinatal outcomes related to GDM (composite of emergency caesarean section delivery, perinatal or neonatal mortality, and infant hospitalization within 28 days). Self-reported via telephone contact post delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Kinra, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (2):
- Indian Institute of Public Health, Hyderabad, India
- MRC/UVRI and LSHTM Uganda Research Unit, Entebbe, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Indian Council of Medical Research guidance stipulates that the main India dataset should be retained in India. Therefore, anonymised data from either country will not made freely available. A controlled access model will be followed: anonymised data will be shared on request, subject to approval from the steering group and Independent Access Advisor. Data sharing will be subject to ethical approval.

REFERENCES:
- [Derived] Birk N, Oakley LL, Mallinson PAC, R D, Babu GR, Nyirenda M, Kinra S. Statistical analysis plan and protocol updates for Gestational diabetes in Uganda and India: Design and Evaluation of Educational Films for Improving Screening and Self-management (GUIDES) trial. Trials. 2023 Aug 12;24(1):520. doi: 10.1186/s13063-023-07508-5. PMID 37568171
- [Derived] Oakley LL, R D, Namara A, Sahu B, Nadal IP, Ana Y, Coombe H, Oteng-Ntim E, Seeley J, Nyirenda M, Babu G, Kinra S. Educational films for improving screening and self-management of gestational diabetes in India and Uganda (GUIDES): study protocol for a cluster-randomised controlled trial. Trials. 2021 Jul 28;22(1):501. doi: 10.1186/s13063-021-05435-x. PMID 34321046